CLINICAL TRIAL: NCT02626767
Title: Effect of Novel High-intensity Interval Training on Cardiometabolic Health and Physical Activity Levels in English Adolescents: A School-based Exploratory Controlled Before-and-after Trial
Brief Title: Effect of Novel High-intensity Interval Training on Health and Fitness Outcomes in English Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Collaborators: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Kathryn Weston, Senior Lecturer in Applied Biosciences for Health, Teesside University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TEES-008/11
Record Dates: First submitted 2015-12-03; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: High-intensity Interval Training
Keywords: high-intensity interval training; adolescents; school-based exercise; cardiometabolic health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants were required to complete a high-intensity interval exercise training intervention, which took place three time per week for 10 weeks. The exercise sessions comprised of 4 to 7 repetitions of 45 s maximal effort exercise, based on boxing, dance, soccer and basketball drills), interspersed with 90-s rest. During each repetitions participants were encouraged to reach >90% of their individual maximal heart rate. Participants were asked to maintain their dietary habits throughout the intervention period.
  Interventions: Other: Novel high-intensity interval exercise training
- Control (No Intervention): Participants were asked to maintain their usual diet, physical education and physical activity habits during the intervention period and were not aware that an exercise intervention was taking place at other study sites.

INTERVENTIONS:
Other: Novel high-intensity interval exercise training — Please see information already included in the 'intervention' arm description.
  Arms: Intervention

SUMMARY:
Low-volume high-intensity interval exercise training may improve aspects of health and fitness in young people, but interventions must be practical and engaging. The investigators examined the effect of a novel school-based low-volume high-intensity interval training programme on health, fitness and physical activity outcomes in adolescent school pupils. 101 English adolescents aged 13-14 years took part in the study. Participants were healthy male and female volunteers, recruited from four schools in Northeast England. Using a non-randomised design, two schools took part in the intervention, and two were assigned to the control. Those in the intervention group completed a 10-week school-based high-intensity interval exercise training programme. The intervention took place three times per week, and comprised of 4-7 repetitions of 45 s maximal effort exercise (boxing, dance, soccer and basketball drills), each interspersed with 90-s rest. Participants were encouraged to work maximally during the 45-s repetitions. Control participants were instructed not to change their lifestyle, dietary or physical activity habits during the intervention period, and maintain their normal school physical education routine. Study outcomes were blood lipid and glucose levels, body composition, cardiorespiratory fitness, carotid intima-media thickness, physical activity levels, serum C-reactive protein levels and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Must attend one of the four schools that the study will take place in
2. Must be in the Year 9 English school year (aged 13-15 years)
3. Must provide parental consent and participant assent
4. Must be free from exclusion criteria

Exclusion Criteria:

1. Symptoms of or known presence of heart disease or major atherosclerotic cardiovascular disease
2. Condition or injury or co-morbidity affecting the ability to undertake exercise
3. Diabetes mellitus
4. Early family history of sudden cardiac death
5. Condition or disorder which is communicable via blood
6. Pregnancy or likelihood of pregnancy

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline (0 weeks) waist circumference at the post-intervention time point (10 weeks) | Baseline (0 weeks) and post-intervention (10-weeks)
Change from baseline (0 weeks) blood lipids at the post-intervention time point (10 weeks) (assessed via finger prick blood sampling) | Baseline (0 weeks) and post-intervention (10-weeks)
Change from baseline (0 weeks) blood glucose at the post-intervention time point (10 weeks) (assessed via finger prick blood sampling) | Baseline (0 weeks) and post-intervention (10-weeks)
Change from baseline (0 weeks) blood pressure at the post-intervention time point (10 weeks) | Baseline (0 weeks) and post-intervention (10-weeks)
Change from baseline (0 weeks) carotid artery intima-media thickness at the post-intervention time point (10 weeks) | Baseline (0 weeks) and post-intervention (10-weeks)
Change from baseline (0 weeks) body mass index at the post-intervention time point (10 weeks) | Baseline (0 weeks) and post-intervention (10-weeks)
Change from baseline (0 weeks) serum C-reactive protein at the post-intervention time point (10 weeks) | Baseline (0 weeks) and post-intervention (10-weeks)
Change from baseline (0 weeks) 20m shuttle run test performance (indirect measure of cardiorespiratory fitness) at the post-intervention time point (10 weeks) | Baseline (0 weeks) and post-intervention (10-weeks)
Change from baseline (0 weeks) daily physical activity levels (assessed via accelerometry) at the post-intervention time point (10 weeks) | Baseline (0 weeks) and post-intervention (10-weeks)
Change from baseline (0 weeks) body weight at the post-intervention time point (10 weeks) | Baseline (0 weeks) and post-intervention (10-weeks)
Change from baseline (0 weeks) percentage body fat at the post-intervention time point (10 weeks) | Baseline (0 weeks) and post-intervention (10-weeks)
Change from baseline (0 weeks) skeletal muscle mass at the post-intervention time point (10 weeks) | Baseline (0 weeks) and post-intervention (10-weeks)

OTHER OUTCOMES:
Heart rate during high-intensity interval training exercise sessions | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L Weston, PhD, Principal Investigator — Teesside University, Middlesbrough,UK

IPD SHARING:
Plan to Share IPD: No
Only group level data will be published from this study.

REFERENCES:
- [Derived] Weston KL, Azevedo LB, Bock S, Weston M, George KP, Batterham AM. Effect of Novel, School-Based High-Intensity Interval Training (HIT) on Cardiometabolic Health in Adolescents: Project FFAB (Fun Fast Activity Blasts) - An Exploratory Controlled Before-And-After Trial. PLoS One. 2016 Aug 3;11(8):e0159116. doi: 10.1371/journal.pone.0159116. eCollection 2016. PMID 27486660